CLINICAL TRIAL: NCT01532518
Title: A Multicenter, Open Label, Ascending 7 Day-Repeated Dose Study to Investigate Efficacy, Safety and Pharmacokinetics of Nepadutant In Infants With Feeding Intolerance
Brief Title: Preliminary Efficacy, Safety and Pharmacokinetics Study of Nepadutant in Infant With Feeding Intolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIC-04
Record Dates: First submitted 2012-01-25; First posted 2012-02-14 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-08

CONDITIONS: Colic
Keywords: Feeding intolerance; Infant; tachykinin antagonist; Infant colic; Nepadutant
MeSH Terms: conditions — Colic | interventions — MEN 11420

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 3 (Experimental): Nepadutant low dose (0.1mg/kg) for 7 days followed by Nepadutant high dose (1mg/kg) for additional 7 days
  Interventions: Drug: Nepadutant
- Cohort 2 (Experimental): Nepadutant medium dose (0.5mg/kg) for 7 days followed by Nepadutant high dose (1mg/kg) for additional 7 days
  Interventions: Drug: Nepadutant
- Cohort 1 (Experimental): Nepadutant low dose (0.1mg/kg) for 7 days followed by Nepadutant medium dose (0.5mg/kg) for additional 7 days
  Interventions: Drug: Nepadutant

INTERVENTIONS:
Drug: Nepadutant — Nepadutant oral solution
  Other Names: MEN 11420

SUMMARY:
The present pilot study is aimed to obtain preliminary data on the effect of three ascending oral dose levels of nepadutant on the relief of symptoms associated with feeding intolerance. In addition, the assessment of drug exposure (PK assessment) will provide additional information on the dose-effect relationship, thus supporting the dose selection and dosing schedule in the future studies.

DETAILED DESCRIPTION:
Feeding intolerance is a transient neuro-developmental phenomenon affecting 25% to 40% of infant and toddler, with a peak at 6 weeks of age. Feeding problems include mainly vomiting, slow feeding, refusal to eat and colic.

Current non pharmacological interventions (e.g. message, restriction in maternal diet in breast-feeding infants) and pharmacological treatments (simethicone, antimuscarinic drugs and antiacids) are largely unsatisfactory.

Nepadutant is postulated to have a therapeutic effect in infant colic since it reverts exaggerated intestinal motility and sensitivity induced by different stimuli through the activation of neurokinin-2 receptors, without interferring on the on physiological gastrointestinal transit.

This phase IIa study is designed to test in each participant infant two out of three oral doses of nepadutant in order to measure its blood levels, safety and efficacy with each dose level to be given for 7 concecutive days.

The experimental clinical phase encompasses the following periods:

* Screening period (no study medication), lasting approximately 7 days prior to randomization
* Treatment period, lasting fourteen days (7 days fore each dose)with once daily administration
* A safety follow-up visit, approximately four weeks after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a clinical diagnosis of feeding intolerance.
* Age ≤ 6 months at the enrolment.
* Normal growth.
* Infants who can refrain from use of erythromycin, metoclopramide, antihistaminic drug, proton pump inhibitors (PPIs), antacids, antimuscarinic drugs, simethicone and dimethicone from 1 week prior randomization until end of study.

Exclusion Criteria:

* Any clinically relevant event (excluding those relevant to the condition under study) which has occurred within one week prior to randomization.
* Any pharmacological treatment starting within one week prior to randomization.
* Infants for whom a change in the diet (i.e. weaning) has been performed within one week prior to randomization or is planned during the study period.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Blumer, MD, PhD, Principal Investigator — The University of Toledo Medical Center 3000 Arlington Avenue, Toledo OH 43614 USA
Locations (5):
- United States (5):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - Kosair Charities Pediatric Clinical Research Unit / University of Louisville, Louisville, Kentucky
  - SUNY Downstate Medical Center, Albany, New York
  - The University of Toledo College of Medicine\The Toledo Children's Hospital, Toledo, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 3 | Cohort 2 | Cohort 1
Started | 6 | 15 | 6
Completed | 6 | 15 | 5
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Infants with Feeding Intolerance
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 3 | Cohort 2 | Cohort 1 | Total
Number analyzed (Participants) | 6 | 15 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Age is in weeks (PGA: post gestational age)
  weeks | 12.52 (4.281) | 13.62 (6.468) | 14.27 (6.559) | 13.52 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 2 | 14
  Male | 2 | 7 | 4 | 13
Race/Ethnicity, Customized [Number; unit: particpants]
  Black or African American | 3 | 4 | 1 | 8
  White | 3 | 8 | 5 | 16
  More than one race | 0 | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 15 | 6 | 27
Weight [Mean (Standard Deviation); unit: Kg] | 5.323 (0.9085) | 5.623 (1.1045) | 5.708 (1.764) | 5.576 (1.1975)
I-GERQ-R total score [Mean (Standard Deviation); unit: Score on a scale] — Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R ), with a minimum-maximum score of 0-42 (minimum for diagnosis >15). The higher values reflect worse outcome. The questionnaire comprised 12 items as questions quantifying aspects of regurgitation (3 questions), crying (3 questions), feeding refusal (2 questions), apnea/cyanosis (2 questions), hiccups and arching. Questions with 4 possible options have a score ranging from 0 to 3; questions with 5 possible options have a score ranging from 0 to 4.
  The scores of each item are summed, so the total score is presented.
  Score on a scale | 24.8 (5.4) | 19 (6.32) | 21.8 (9.91) | 20.8 (7.22)

OUTCOME MEASURES:

1. Primary Outcome: The Absolute Differences of I-GERQ-R Total Score at V3 (End of First Week of Treatment) Respect to the Baseline (V2).
Description: Results obtained at V2 serve as baseline values for the assessment of effects at V3 (i.e. end of first week of treatment).
  Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R ), with a minimum-maximum score of 0-42 (minimum for diagnosis >15). The higher values reflect worse outcome. The questionnaire comprised 12 items as questions quantifying aspects of regurgitation (3 questions), crying (3 questions), feeding refusal (2 questions), apnea/cyanosis (2 questions), hiccups and arching. Questions with 4 possible options have a score ranging from 0 to 3; questions with 5 possible options have a score ranging from 0 to 4.
  The scores of each item are summed, so the total score is presented.
Time Frame: Baseline (V2) and end of first week of treatment (V3)
Population: Infants with feeding intolerance who received at least 1 dose of nepadutant. In the 3rd cohort 1 subject didn't report I-GERQ-R score at randomization. In the 1rst cohort 1 patient early terminated after V2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 3 | Cohort 2 | Cohort 1
Number analyzed (Participants) | 5 | 15 | 5
score on a scale | -6.8 (9.55) | -7.6 (5.5) | -6.8 (5.81)

2. Primary Outcome: The Absolute Differences of I-GERQ-R Total Score at V4 (End of 2nd Week of Treatment) Respect to V3 (End of 1st Week of Treatment).
Description: The results obtained at V3 are used as baseline for the second week treatment period (V4).
  Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R ), with a minimum-maximum score of 0-42 (minimum for diagnosis >15). The higher values reflect worse outcome. The questionnaire comprised 12 items as questions quantifying aspects of regurgitation (3 questions), crying (3 questions), feeding refusal (2 questions), apnea/cyanosis (2 questions), hiccups and arching. Questions with 4 possible options have a score ranging from 0 to 3; questions with 5 possible options have a score ranging from 0 to 4.
  The scores of each item are summed, so the total score is presented.
Time Frame: V3 (end of 1st week of treatment) and V4 (end of 2nd week of treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score as sum of units
Arm/Group | Cohort 3 | Cohort 2 | Cohort 1
Number analyzed (Participants) | 5 | 15 | 5
Score as sum of units | -15.2 (5.54) | -11.9 (6.8) | -8.6 (6.66)

3. Primary Outcome: The Absolute Differences of I-GERQ-R Total Score at V5 (Follow-up) Respect to V2 (Baseline).
Description: Results obtained at V2 serve as baseline values for follow-up assessment 2 weeks after the last administered dose (V5) Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R ), with a minimum-maximum score of 0-42 (minimum for diagnosis >15). The higher values reflect worse outcome. The questionnaire comprised 12 items as questions quantifying aspects of regurgitation (3 questions), crying (3 questions), feeding refusal (2 questions), apnea/cyanosis (2 questions), hiccups and arching. Questions with 4 possible options have a score ranging from 0 to 3; questions with 5 possible options have a score ranging from 0 to 4.
  The scores of each item are summed, so the total score is presented.
Time Frame: Baseline (V2) and follow up 2 weeks after the last administered dose (V5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score as sum of units
Arm/Group | Cohort 3 | Cohort 2 | Cohort 1
Number analyzed (Participants) | 5 | 15 | 5
Score as sum of units | -7.8 (7.6) | -11.1 (6.78) | -9.8 (7.4)

4. Primary Outcome: I-GERQ-R Score Changes vs Baseline (Visit 2) by First Dose Level (0.1mg/kg and 0.5mg/kg).
Description: Change in Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R) Score. Assessing the I-GERQ-R score changes vs baseline (Visit 2) by first dose level (0.1mg/kg and 0.5mg/kg). Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R ), with a minimum-maximum score of 0-42 (minimum for diagnosis >15). The higher values reflect worse outcome. The questionnaire comprised 12 items as questions quantifying aspects of regurgitation (3 questions), crying (3 questions), feeding refusal (2 questions), apnea/cyanosis (2 questions), hiccups and arching. Questions with 4 possible options have a score ranging from 0 to 3; questions with 5 possible options have a score ranging from 0 to 4.
  The scores of each item are summed, so the total score is presented.
Time Frame: Baseline (V2) and end of 1st week of treatment(V3)
Population: Subjects with feeding intolerance who received at least 1 dose of nepadutant (first dose level 0.1mg/kg and 0.5 mg/kg).
  One subject in the 3rd cohort didn't report I-GERQ-R score at V2.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Low Dose Level (0.1mg/kg): Subjects who received at least 1 dose of nepadutant 0.1mg/kg
- Medium Dose Level 0.5mg/kg: Subjects who received at least 1 dose of nepadutant 0.5mg/kg
Arm/Group | Low Dose Level (0.1mg/kg) | Medium Dose Level 0.5mg/kg
Number analyzed (Participants) | 10 | 15
score on a scale | -6.8 (7.31) | -7.6 (5.5)

5. Primary Outcome: I-GERQ-R Score Changes vs Visit 3 by Second Dose Level (0.5mg/kg and 1mg/kg).
Description: Change in Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R) Score. Assessing the I-GERQ-R score changes vs Visit 3 by second dose level (0.5mg/kg and 1mg/kg).
  Infant Gastroesophageal Reflux Questionnaire Revised (I-GERQ-R ), with a minimum-maximum score of 0-42 (minimum for diagnosis >15). The higher values reflect worse outcome. The questionnaire comprised 12 items as questions quantifying aspects of regurgitation (3 questions), crying (3 questions), feeding refusal (2 questions), apnea/cyanosis (2 questions), hiccups and arching. Questions with 4 possible options have a score ranging from 0 to 3; questions with 5 possible options have a score ranging from 0 to 4.
  The scores of each item are summed, so the total score is presented.
Time Frame: end of first week of treatment (V3) and end of second week of treatment (V4)
Population: Subjects with feeding intolerance who received at least 1 dose of nepadutant (second dose level 0.5mg/kg and 1 mg/kg)
  1 subject in the first cohort early terminated after V2
Measure: Mean (Standard Deviation); unit: Score as sum of units
Groups:
- Medium Dose Level (0.5mg/kg): Subjects who received at least 1 dose of nepadutant 0.5mg/kg
- High Dose Level 1mg/kg: Subjects who received at least 1 dose of nepadutant 1mg/kg
Arm/Group | Medium Dose Level (0.5mg/kg) | High Dose Level 1mg/kg
Number analyzed (Participants) | 5 | 21
Score as sum of units | -1.4 (0.89) | -4.9 (4.41)

6. Secondary Outcome: Incidence and Severity of AEs_ Number of Adverse Events by Treatment Dose Level
Description: The analysis is by treatment - Each infant was treated with two out of three ascending dose (0.1, 0.5 or 1.0 mg/kg), therefore counted in more than one dose level.
Time Frame: up to 4 weeks
Population: All subjects who received at least one administration of study treatment including dose tolerability test (safety population)
Measure: Number; unit: Number of events
Groups:
- High Dose Level (1.0 mg/Kg): Subjects who received at least 1 dose of nepadutant 1.0mg/kg (Subjects who took Nepadutant 1.0 mg/dl for the additional 7 days - coming from Nepadutant 0.1 mg/kg and 0.5 mg/kg)
  Nepadutant: Nepadutant oral solution
- Medium Dose Level (0.5mg/Kg): Subjects who received at least 1 dose of nepadutant 0.5 mg/kg (subjects who took Nepadutant 0.5 mg/dl for the first 7 days AND subjects who took Nepadutant 0.5 mg/dl for the additional 7 days - coming from Neapdutant 0.1 mg/kg)
  Nepadutant: Nepadutant oral solution
- Low Dose Level(0.1mg/Kg): Subjects who received at least 1 dose of nepadutant 0.1 mg/kg (subjects who took Nepadutant 0.1mg/dl for the first 7 days)
  Nepadutant: Nepadutant oral solution
Arm/Group | High Dose Level (1.0 mg/Kg) | Medium Dose Level (0.5mg/Kg) | Low Dose Level(0.1mg/Kg)
Number analyzed (Participants) | 21 | 21 | 12
Number of events
  gastrointestinal disorder | 6 | 4 | 3
  General disorders and administration site conditio | 1 | 0 | 0
  Infections and infestations | 7 | 2 | 1
  Injury, poisoning and procedural complications | 1 | 1 | 0
  Psychiatric disorders | 0 | 0 | 1
  Respiratory, thoracic and medistinal disorders | 3 | 1 | 1
  Skin and subcutaneous tissue disorders | 3 | 1 | 3

7. Secondary Outcome: A Population Pharmacokinetic Analysis to Characterize the Plasma Concentration-time Course for Nepadutant in Infant With Colics From NIC-04
Description: The population pharmacokinetic analyses is presented. PopPK Clearance estimated with a one compartment model with first order absorption and elimination.
Time Frame: 0.5, 1, 2, 3 hours post Single Dose and 24 hours post Repeated Dose
Population: At visit 2, samples from 12 subjects in 0.1 mg/kg and from 15 subjects in 0.5 mg/kg.
  At visit 3*, 4*: samples from 15 subjects in 0.1 - 0.5 mg/kg cohort, from 5 in 0.5 - 1 mg/kg cohort and from 6 in 0.1 - 1 mg/kg cohort.
  *N=26 instead of 27 as one patient early terminated the study
Measure: Mean (95% Confidence Interval); unit: L/h
Arm/Group | Cohort1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 6 | 15 | 6
L/h | 1.24 [0.919 to 1.57] | 1.31 [1.03 to 1.59] | 1.64 [1.39 to 1.89]

8. Secondary Outcome: A Population Pharmacokinetic Analysis to Characterize the Plasma Concentration-time Course for Nepadutant in Infant With Colics From NIC-04
Description: PopPK Volume estimated with a one compartment model with first order absorption and elimination. NOTE: for this measure, no inter-individual variability was estimated, therefore the value for each cohort corresponds to the typical value.
Time Frame: 0.5, 1, 2, 3 hours post Single Dose and 24 hours post Repeated Dose
Population: At visit 2, samples from 6 subjects in Cohort 1 at 0.1mg/kg; 6 subjects in Cohort 3 at 0,1 mg/kg; 15 subjects in Cohort 2 at 0.5 mg/kg.
  At visit 3*, 4*: samples from 5 subjects in Cohort 1 (0.1 - 0.5 mg/kg), 15 subjects in Cohort 2 (0.5 - 1 mg/kg) and 6 subjects in Cohort 3 (0.1 - 1 mg/kg).
Measure: Mean (Full Range); unit: L
Groups:
- Cohort 1, 2, and 3: Overall population participating to the study for PoP PK analysis
Arm/Group | Cohort 1, 2, and 3
Number analyzed (Participants) | 27
L | 22.5 [NA to NA] — no inter-individual variability was estimated, the value for all cohorts corresponds to the typical value.

9. Secondary Outcome: A Population Pharmacokinetic Analysis to Characterize the Plasma Concentration-time Course for Nepadutant in Infant With Colics From NIC-04
Description: The population pharmacokinetic analyses is presented. PopPK Ka estimated with a one compartment model with first order absorption and elimination. NOTE: for this measure, no inter-individual variability was estimated, therefore the value for each cohort corresponds to the typical value.
Time Frame: 0.5, 1, 2, 3 hours post Single Dose and 24 hours post Repeated Dose
Population: as for outcome 8
Measure: Mean (Full Range); unit: 1/h
Groups:
- Cohort 1, 2 and 3: Data from the 3 cohorts used for PoP PK analysis
Arm/Group | Cohort 1, 2 and 3
Number analyzed (Participants) | 27
1/h | 206 [NA to NA] — no inter-individual variability was estimated, therefore the value for each cohort corresponds to the typical value.

10. Secondary Outcome: A Population Pharmacokinetic Analysis to Characterize the Plasma Concentration-time Course for Nepadutant in Infant With Colics From NIC-04
Description: The population pharmacokinetic analyses is presented. The PopPK parameter fraction of the dose absorbed (F1) is estimated with a one compartment model with first order absorption and elimination.The results are presented fraction of the absorbed dose with 95% CI of the parameter estimate value
Time Frame: 0.5, 1, 2, 3 hours post Single Dose and 24 hours post Repeated Dose
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: fraction of dose absorbed
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 6 | 15 | 6
fraction of dose absorbed | 0.0275 [0.0199 to 0.0352] | 0.0342 [0.0250 to 0.0433] | 0.0346 [0.0346 to 0.0377]

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Analysed for the Safety Population (all patients who received the study drug) The analysis is by treatment - Each infant was treated with two out of three ascending dose (0.1, 0.5 or 1.0 mg/kg), therefore counted in more than one dose level.
Arm/Group | High Dose Level (1.0 mg/Kg) | Medium Dose Level (0.5mg/Kg) | Low Dose Level(0.1mg/Kg)
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/21 | 1/12
Other Adverse Events (participants affected / at risk) | 12/21 | 2/21 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Level (1.0 mg/Kg) (N=21) | Medium Dose Level (0.5mg/Kg) (N=21) | Low Dose Level(0.1mg/Kg) (N=12)
Hospitalisation for investigation for suspected seizures (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — 10 wks-old male-familiar history of seizure disorders.It started 6days after the last drug intake (nepadutant 0.1mg/kg early terminate after 3drug intakes).It reported as "moderate","not related" to nepadutant by investigator. It resolved: no sequel.
Laryngeal Edema-post intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Prolongation of hospitalization due to post-intubation laryngeal edema in a 22wks-old female.It started 4days after the end of the 2weeks of treatment:it reported as "moderate","not related" to the treatment by investigators.It resolved:no sequel.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Level (1.0 mg/Kg) (N=21) | Medium Dose Level (0.5mg/Kg) (N=21) | Low Dose Level(0.1mg/Kg) (N=12)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Teething (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Screaming (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory atract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seborrhoic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study performed in a small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The results of the study cannot be submitted for presentation, abstract, poster exhibition, or publication by the investigator until Menarini Ricerche S.p.A.

has reviewed/commented and agreed to any publication.